CLINICAL TRIAL: NCT00911027
Title: A Phase III Study to Compare SonoVue Guided Prostate Biopsy With Systematic Biopsy in the Detection of Prostate Malignant Lesions in Patients With Suspected Prostate Cancer
Brief Title: SonoVue Guided Prostate Biopsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure to meet primary objective
Sponsor: Bracco Diagnostics, Inc (Industry)
Collaborators: Bracco Imaging S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BR1-127
Record Dates: First submitted 2009-05-07; First posted 2009-06-01 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Biopsy; Guided; Contrast; Enhanced; SonoVue; Suspicion of prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SonoVue guided biopsy (Experimental)
  Interventions: Drug: Contrast-enhanced ultrasound guided biopsy
- Systematic biopsy (Other)
  Interventions: Procedure: ultrasound guided systematic biopsy

INTERVENTIONS:
Drug: Contrast-enhanced ultrasound guided biopsy — One to two bolus (each 2.4mL) of SonoVue per patient in the optimization part
  One to four bolus (each 2.4mL) of SonoVue per patient in the main part
  Other Names: SonoVue guided biopsy
  Arms: SonoVue guided biopsy
Procedure: ultrasound guided systematic biopsy — Current practice of ultrasound guided systematic biopsy
  Arms: Systematic biopsy

SUMMARY:
This is a phase III European multicenter, open label, prospective study to assess the diagnostic accuracy of the use of SonoVue contrast agent to guide prostate biopsies in comparison with the current practice of ultrasound guided systematic biopsy. The trial will involve 15-20 European Centers.

ELIGIBILITY:
Inclusion Criteria:

* Male patient, age ≥ 40 years old
* Optimization part only: Diagnosis of prostate cancer
* Main part: Suspected prostate cancer scheduled for first biopsy and tPSA ≤ 10 ng/mL OR already submitted to one systematic bioptic procedure with negative results currently under follow up procedure due to a persistent indication.
* Written Informed Consent and willing to comply with protocol requirements

Exclusion Criteria:

* Documented acute prostatitis or urinary tract infections
* Known allergy to sulphur hexafluoride micro bubbles
* Any clinically unstable cardiac condition within 7 days prior to SonoVue® administration such as:
* evolving or ongoing myocardial infarction
* typical angina at rest within the previous 7 days
* significant worsening of cardiac symptoms within the previous 7 days
* recent coronary artery intervention or other factors suggesting clinical instability (e.g., recent deterioration of ECG, laboratory or clinical findings)
* acute cardiac failure, class III/IV cardiac failure
* severe cardiac rhythm disorders
* right-to-left shunts
* Severe pulmonary hypertension or uncontrolled systemic hypertension or respiratory distress syndrome
* Bioptic procedure within 30 days before admission into this study (this exclusion criterion is only for the main part of the study)
* Determined by the Investigator that the patient is clinically unsuitable for the study
* Participation in a concurrent clinical trial or in another trial within the past 30 days
* Repeated participation in this trial (the patient should not be enrolled twice in the present study)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Determination of potentiality of SonoVue to guide prostate biopsy increasing detection rate of malignant lesions of 6% points (absolute terms) compared to detection rate of conventional systematic biopsy on patients candidates to a bioptic procedure. | Day 1

SECONDARY OUTCOMES:
Evaluation of the rate of patients negative to the systematic biopsy among the population that will not receive the targeted biopsy | Day 1
Assessment of potentiality of SonoVue guided biopsy to increase % of positive bioptic cores compared to % of positive cores obtained with systematic biopsy, intra-patient in the population of the patients that received both bioptic procedures. | Day 1
Evaluation of the Gleason Score of bioptic samples and its relationship with the contrast enhanced signal assessment scores. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Storto, MD, Study Chair — Bracco Diagnostics, Inc
Locations (17):
- Medical University Innsbruck, Innsbruck, Austria
- University Hospital K.U. Leuven, Leuven, Belgium
- France (3):
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Necker-Enfants Malades, Paris
  - CHRU Tours - Hôpital Bretonneau, Tours
- Germany (3):
  - Institut für Radiologie der Charité, Berlin
  - Martini-Klinik, Prostate Cancer Center, Hamburg
  - Urologische Klinik und Poliklinik, Munich
- Italy (6):
  - Orsola-Malpighi Hospital, Urology and Radiology Unit "Malpighi", Bologna
  - Ospedale Valduce, Como
  - European Institute of Oncology, Milan
  - I.R.C.C.S. San Raffaele, Milan
  - University of Palermo, Palermo
  - University of Trieste, Trieste
- Netherlands (2):
  - AMC University Amsterdam, Amsterdam
  - Erasmus MC, Rotterdam
- Imperial College NHS Trust - Charing Cross, London, United Kingdom